CLINICAL TRIAL: NCT00702507
Title: Prospective 2-Year Longitudinal Study to Assess for Miconazole Resistance in Candida Spp. With Repeated Treatment Courses of 0.25% Miconazole Nitrate Ointment in Neonates and Infants up to 1 Year of Age With Recurrent Moderate-Severe Diaper Dermatitis Complicated by Cutaneous Candidiasis
Brief Title: Prospective Two-Year Study to Assess Miconazole Nitrate Resistance in Neonates and Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114678; BT0100-402-USA (Other: Barrier Therapeutics)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Diaper Rash
Keywords: Diaper dermatitis complicated by candidiasis
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miconazole Nitrate (Active Comparator)
  Interventions: Drug: 0.25 % Miconazole Nitrate Ointment

INTERVENTIONS:
Drug: 0.25 % Miconazole Nitrate Ointment — Topical Application
  Other Names: Vusion

SUMMARY:
The purpose of this study is to determine whether repeated use of 0.25% miconazole nitrate ointment in newborns and infants with a yeast infection in the diaper area causes the yeast to become resistant to the drug.

DETAILED DESCRIPTION:
The objective of this study is to investigate the potential for the development of resistance in Candida spp. after repeated treatment courses of 0.25% miconazole nitrate ointment in neonates and infants up to one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female neonate or infant up to 1 year of age with Fitzpatrick Skin Type I-VI
* Clinical evidence of diaper dermatitis and a positive KOH result for pseudohyphae and/or budding yeast at baseline visit
* Overall Diaper Dermatitis Severity Index score at baseline visit of 4-8 (must include an overall clinical grade of at least 2 for erythema)
* Wear commercially available diapers day and night for at least 7 days prior to enrollment and during the course of the 2 year study
* Caretaker must complete informed consent process

Exclusion Criteria:

* Known sensitivity to any component of the formulation
* No other skin conditions that may confound the evaluation of the drug efficacy or tolerability
* Known sensitivity to skin care toiletry products or diapers
* History of HIV positive
* Chronic illnesses that require systemic medication that may confound the evaluation of study drug efficacy or tolerability (antibiotic therapy is not included)
* Treatment with a prescription product for diaper dermatitis or other skin condition 7 days prior to enrollment

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - Sheila Fallon Friedlander, MD, San Diego, California
  - David Rodriguez, MD, Coral Gables, Florida
  - Lawrence Schachner, MD, Miami, Florida
  - Wilson P. Andrews Jr., MD, Marietta, Georgia
  - Lewis Purnell, MD, San Antonio, Texas
- Daisy Blanco, MD, Santo Domingo, Dominican Republic
- Manuel Briones, MD, Guayaquil, Ecuador
- Zila Espinosa, MD, Panama City, Panama

REFERENCES:
- [Derived] Blanco D, van Rossem K. A prospective two-year assessment of miconazole resistance in Candida spp. With repeated treatment with 0.25% miconazole nitrate ointment in neonates and infants with moderate to severe diaper dermatitis complicated by cutaneous candidiasis. Pediatr Dermatol. 2013 Nov-Dec;30(6):717-24. doi: 10.1111/pde.12107. Epub 2013 May 16. PMID 23675632

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 phases: initial treatment phase (14-day study period) and a follow-up phase (2-year study period).
Groups:
- Vusion Treatment: Participants were treated with Vusion ointment containing 0.25 percent miconazole nitrate for 7 days. A follow-up post-treatment visit was conducted at Study Day 14. Further, participants were followed for 2 years. If there was a recurrent episode of diaper dermatitis complicated by candidiasis (DDCC) during the 2-year follow-up period, the participant was treated for 7 days with Vusion ointment.
Period: Initial Treatment Phase
Arm/Group | Vusion Treatment
Started | 200
Completed | 159
Not Completed | 41
Not completed — Adverse Event | 2
Not completed — Participant's Caretaker Withdrew Consent | 3
Not completed — Lost to Follow-up | 2
Not completed — Negative Candida Culture | 34
Period: Follow-up Phase
Arm/Group | Vusion Treatment
Started | 159
Completed | 132
Not Completed | 27
Not completed — Participant's Caretaker Withdrew Consent | 1
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 23
Not completed — Late Enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 200
Age Continuous [Mean (Standard Deviation); unit: Months] | 6.6 (3.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 88
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40
  Black | 17
  Hispanic/Latino | 121
  Hispanic/Persian | 1
  Hispanic/White | 5
  White/Black | 1
  Multiracial | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Cure (OC)
Description: OC was defined as both clinical (therapeutic) cure with total resolution of signs/symptoms (no clinical signs of infection) and microbiological cure with mycological eradication (both negative potassium hydroxide [KOH] and culture results). Participants who had OC were categorized as "Successes"; those without OC were categorized as "Failures." Any discontinued or lost to follow-up participant was also considered a failure.
Time Frame: Test-of-cure visit (Day 14) of initial treatment episode
Population: Modified Intent-to-Treat (MITT) Population: all participants who were dispensed study drug and had demonstrated clinical symptoms of diaper dermatitis (DD) (DD severity index score of 4-8; clinical erythema grade of >=2 [see outcome measure #4 for a description]) and confirmed Candida species (positive baseline KOH and culture for Candida species)
Measure: Number; unit: participants
Groups:
- Vusion Treatment: Participants were treated with Vusion ointment containing 0.25 percent miconazole nitrate for 7 days. A follow-up post-treatment visit was conducted at Study Day 14. Further, participants were followed for 2 years. If there was a recurrent episode of DDCC during the 2-year follow-up period, the participant was treated for 7 days with Vusion ointment.
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 168
participants
  Success | 49
  Failure | 119
Statistical Analysis 1: Comparison: Vusion Treatment; Test type: Superiority or Other; Percentage of participants = 29.2, 95% CI 2-sided [22.4 to 36.7] — Percentage of participants with overall cure at the test-of-cure visit (Day 14) of the initial episode for participants in the MITT Population

2. Secondary Outcome: Number of Participants With Clinical Cure
Description: Participants were evaluated for clinical cure, which was defined as therapeutic cure with total resolution of signs and symptoms (i.e., no clinical signs of infection). Participants who had clinical cure were categorized as "Successes"; those without clianical cure were categorized as "Failures." Any discontinued or lost to follow-up participant was also considered a failure.
Time Frame: Test-of-cure visit (Day 14) of initial treatment episode
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 168
participants
  Success | 83
  Failure | 85

3. Secondary Outcome: Number of Participants With Mycological Cure
Description: Participants were evaluated for mycological cure, which was defined as mycological eradication with negative KOH and culture results. Participants who had mycological cure were categorized as "Successes"; those without mycological cure were categorized as "Failures." Any discontinued or lost to follow-up participant was also considered a failure.
Time Frame: Test-of-cure visit (Day 14) of initial treatment episode
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 168
participants
  Success | 77
  Failure | 91

4. Secondary Outcome: Clinical Evaluations Using the Diaper Dermatitis Severity Index Score for Initial Treatment Episode
Description: The diaper dermatitis severity index score was calculated as the sum of severity grades for each parameter evaluated (erythema, papules or pustules, and erosions) for the initial treatment episode. The maximum score possible for the diaper dermatitis severity index is 8. Rating scale for Erythema: 0 (none to trace), 1 (mild [pink]), 2 (moderate [red]), 3 (severe [beefy red]). Rating scale for Papules or Pustules: 0 (none to trace [0]), 1 (few [1-10]), 2 (multiple [11-20]), 3 (many [21-40]), 4 (abundant [more than 40]. Rating scale for Erosions: 0 (absent), 1 (present).
Time Frame: Test-of-cure visit (Day 14) of initial treatment episode
Population: MITT Population. Participants with missing data were not included in this analysis.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 160
scores on a scale | 0.0 [0 to 7]

5. Secondary Outcome: Clinical Evaluations Using Change From Baseline in the Dermatitis Severity Index Score at Day 14 of the Initial Treatment Episode
Description: The diaper dermatitis severity index score was calculated as the sum of severity grades for each parameter evaluated (erythema, papules or pustules, and erosions). Change from baseline=baseline value minus Day 14 value. The maximum score possible for the diaper dermatitis severity index is 8. Rating scale for Erythema: 0 (none to trace), 1 (mild [pink]), 2 (moderate [red]), 3 (severe [beefy red]). Rating scale for Papules or Pustules: 0 (none to trace [0]), 1 (few [1-10]), 2 (multiple [11-20]), 3 (many [21-40]), 4 (abundant [more than 40]. Rating scale for Erosions: 0 (absent), 1 (present).
Time Frame: Test-of-cure visit (Day 14) of initial treatment episode
Population: MITT Population. Participants with missing data were not included in this analysis.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 160
scores on a scale | -5.0 [-8 to 1]

6. Secondary Outcome: Number of Participants With Overall Cure (OC) of First to Third Recurrent Episodes (RE)
Description: OC was defined as both clinical (therapeutic) cure with total resolution of signs/symptoms (no clinical signs of infection) and microbiological cure with mycological eradication (both negative potassium hydroxide and culture results) at TOC visit for initial episode (ep.) to third ep. Participants (par) who had OC were categorized as "Successes"; those without OC were categorized as "Failures" (discontinued/lost to follow-up par were also failures). A RE is not temporally associated with a prior episode (PE) irrespective of whether the PE involves continuing treatment with study medication.
Time Frame: Test-of-cure (TOC) visit (Day 14) of first to third recurrent episodes (up to approximately 1 year and 7 months)
Population: MITT Population: only those participants with confirmed recurrence were analyzed
Measure: Number; unit: participants
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 35
participants
  First Recurrence, Success; n=35 | 11
  First Recurrence, Failure; n=35 | 24
  Second Recurrence, Success; n=10 | 5
  Second Recurrence, Failure; n=10 | 5
  Third Recurrence, Success; n=4 | 2
  Third Recurrence Failure; n=4 | 2

7. Secondary Outcome: Number of Participants With Clinical Cure of First to Third Recurrent Episodes
Description: Participants were evaluated for clinical cure, which was defined as therapeutic cure with total resolution of signs and symptoms (i.e., no clinical signs of infection). Participants who had clinical cure were categorized as "Successes"; those without clinical cure were categorized as "Failures." Any discontinued or lost to follow-up participant was also considered a failure.
Time Frame: Test-of-cure visit (Day 14) of first to third recurrent episodes (up to approximately 1 year and 7 months)
Population: MITT Population: only those participants with confirmed recurrence were analyzed
Measure: Number; unit: participants
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 35
participants
  First Recurrence, Success; n=35 | 20
  First Recurrence, Failure; n=35 | 15
  Second Recurrence, Success; n=10 | 5
  Second Recurrence, Failure; n=10 | 5
  Third Recurrence, Success; n=4 | 3
  Third Recurrence Failure; n=4 | 1

8. Secondary Outcome: Number of Participants With Mycological Cure of First to Third Recurrent Episodes
Description: as for outcome 3
Time Frame: Test-of-cure visit (Day 14) of first to third recurrent episodes (up to approximately 1 year and 7 months)
Population: MITT Population: only those participants with confirmed recurrence were analyzed
Measure: Number; unit: participants
Arm/Group | Vusion Treatment
Number analyzed (Participants) | 35
participants
  First Recurrence, Success; n=35 | 16
  First Recurrence, Failure; n=35 | 19
  Second Recurrence, Success; n=10 | 7
  Second Recurrence, Failure; n=10 | 3
  Third Recurrence, Success; n=4 | 3
  Third Recurrence Failure; n=4 | 1

ADVERSE EVENTS:
Groups:
- Vusion Initial Treatment Phase: Participants were treated with Vusion ointment containing 0.25 percent miconazole nitrate for 7 days. A follow-up post-treatment visit was conducted at Study Day 14.
- Vusion Follow-up Phase: After the Initial Treatment Phase participants were followed for 2 years. If there was a recurrent episode of diaper dermatitis complicated by candidiasis (DDCC) during the 2-year follow-up period, the participant was treated for 7 days with Vusion ointment containing 0.25 percent miconazole nitrate.
Arm/Group | Vusion Initial Treatment Phase | Vusion Follow-up Phase
Serious Adverse Events (participants affected / at risk) | 0/200 | 3/168
Other Adverse Events (participants affected / at risk) | 42/200 | 133/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vusion Initial Treatment Phase (N=200) | Vusion Follow-up Phase (N=168)
Febrile Convulsion (Nervous system disorders) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vusion Initial Treatment Phase (N=200) | Vusion Follow-up Phase (N=168)
Conjunctivitis (Eye disorders) | 1 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 41
Vomiting (Gastrointestinal disorders) | 3 | 22
Pyrexia (General disorders) | 18 | 79
Amoebiasis (Infections and infestations) | 0 | 8
Bronchitis (Infections and infestations) | 1 | 11
Diarrhoea infectious (Infections and infestations) | 0 | 9
Ear infection (Infections and infestations) | 2 | 11
Impetigo (Infections and infestations) | 2 | 8
Influenza (Infections and infestations) | 2 | 7
Nasopharyngitis (Infections and infestations) | 19 | 69
Otitis media acute (Infections and infestations) | 2 | 13
Pharyngitis (Infections and infestations) | 0 | 12
Pharyngotonsilitis (Infections and infestations) | 0 | 15
Respiratory tract infection (Infections and infestations) | 0 | 10
Rhinitis (Infections and infestations) | 2 | 14
Tonsillitis (Infections and infestations) | 1 | 28
Varicella (Infections and infestations) | 0 | 6
Viral infection (Infections and infestations) | 1 | 10
Viral rash (Infections and infestations) | 3 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 26
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.